CLINICAL TRIAL: NCT05519930
Title: Pancreatic Cancer Early Detection Registry
Status: Completed | Type: Observational
Sponsor: Hoag Memorial Hospital Presbyterian (Other)
Responsible Party: Sponsor
Other Study IDs: 113-16-CA
Record Dates: First submitted 2022-08-22; First posted 2022-08-29 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic Cancer; Hereditary High Risk
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 99 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: hereditary high risk pancreatic cancer — Data collection trial for hereditary high risk pancreatic cancer patients.

SUMMARY:
Identify individuals who are at moderate and high risk or predisposed to developing pancreatic cancer with a familial history in which data collected from this study will be used to identify clinical factors associated with early detection of pancreatic cancer.

DETAILED DESCRIPTION:
Pancreatic cancer is the fourth leading cause of cancer death in both men and women in the United States. In 2015, there were 49,000 new diagnoses with 41,000 deaths . A recent analysis of the pedigrees in the National Familial Pancreatic Tumor Registry found that individuals with a family history of pancreatic cancer in first-degree relatives are at an increased risk of developing pancreatic cancer themselves. There are more than a dozen inherited germline mutations that increase the risk of pancreatic cancer in these family members. In an attempt to lower the number of individuals that develop advanced pancreatic cancer, an early-detection program is created to detect tumors at a stage early enough that treatment is likely to be successful. Numerous treatment options exist such as surveillance, radiation therapy, systemic therapy and surgery. Determining which treatment option will be implemented is based on the stage and grade of the tumor/cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Eligible subjects must be ≥ 18 years of age
2. Meet one of the following criteria:

   * All affected on the same side of the family (maternal/paternal) unless otherwise specified FDR = first degree relative (parent, sibling, child)
   * SDR = second degree relative (e.g., aunt, uncle, grandparent, half-sibling, niece and nephew)
   * TDR = third degree relative (e.g., cousin, half-aunt or half-uncle)

     * 1 FDR with pancreatic cancer < age 55

       -≥2 FDR, SDR or TDR with pancreatic cancer at any age
     * Genetic syndrome with pancreatic cancer
     * FDR or SDR with pancreatic cancer at any age and Ashkenazi ancestry
     * FDR or SDR with pancreatic cancer at any age and:

       * 1 relative with ovarian cancer at any age or
       * 1 relative with breast cancer ≤50 or
       * 2 relatives with breast, pancreatic or prostate cancer (Gleason score ≥7) at any age
     * Family history of melanoma OR
     * Has previously had genetic testing and has been determined to have a pathogenic gene variant.
     * FDR with a pathogenic gene variant

Exclusion Criteria:

1. Prior treatment of pancreatic cancer including radiation therapy, systemic therapy and/or surgery.
2. Current treatment of pancreatic cancer including radiation therapy, systemic therapy and/or surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 2. Meet one of the following criteria:
  * All affected on the same side of the family (maternal/paternal) unless otherwise specified FDR = first degree relative (parent, sibling, child)
  * SDR = second degree relative (e.g., aunt, uncle, grandparent, half-sibling, niece and nephew)
  * TDR = third degree relative (e.g., cousin, half-aunt or half-uncle)
    * 1 FDR with pancreatic cancer < age 55
      -≥2 FDR, SDR or TDR with pancreatic cancer at any age
    * Genetic syndrome with pancreatic cancer
    * FDR or SDR with pancreatic cancer at any age and Ashkenazi ancestry
    * FDR or SDR with pancreatic cancer at any age and:
      * 1 relative with ovarian cancer at any age or
      * 1 relative with breast cancer ≤50 or
      * 2 relatives with breast, pancreatic or prostate cancer (Gleason score ≥7) at any age
    * Family history of melanoma OR
    * Has previously had genetic testing and has been determined to have a pathogenic gene variant.
    * FDR with a pathogenic gene variant
Sampling Method: Probability Sample
Enrollment: 326 (Actual)
Dates: Start 2016-10-18 (Actual); Primary Completion 2023-07-27 (Actual); Study Completion 2023-07-27 (Actual)

PRIMARY OUTCOMES:
Evaluation of imaging for early detection of pancreatic cancer in the high-risk group as defined by inclusion criteria to determine their level of risk and perform surveillance accordingly. | Eight years
  Imaging includes CT/MRI abdomen with and without contrast using the pancreatic protocol, screening for solid pancreatic lesions, atypical cysts and IPMN, pancreatic duct dilatation, pancreas divisum.
Evaluation of blood samples for early detection of pancreatic cancer in the high-risk group as defined by inclusion criteria to determine their level of risk and perform surveillance accordingly. | Eight years
Evaluation of endoscopic ultrasound for early detection of pancreatic cancer in the high-risk group as defined by inclusion criteria to determine their level of risk and perform surveillance accordingly | Eight years

CONTACTS AND LOCATIONS:
Overall Officials: Valentina Dalili-Shoaie, MD, Principal Investigator — Hoag Memorial Hospital Presbyterian
Locations (1):
- Hoag Memorial Hospital Presbyterian, Newport Beach, California, United States

IPD SHARING:
Plan to Share IPD: No